CLINICAL TRIAL: NCT03748680
Title: Implementing Non-invasive Circulating Tumor DNA Analysis to Optimize the Operative and Postoperative Treatment for Patients With Colorectal Cancer
Brief Title: IMPROVE Intervention Trial Implementing Non-invasive Circulating Tumor DNA Analysis to Optimize the Operative and Postoperative Treatment for Patients With Colorectal Cancer
Acronym: IMPROVE-IT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karen-Lise Garm Spindler (Other)
Responsible Party: Sponsor-Investigator, Karen-Lise Garm Spindler, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFE-1803
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Cancer; Circulating Tumor DNA; Adjuvant Chemotherapy; Progression Free Survival
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: A open label 1:1 randomized phase II exploratory study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Active Comparator): Intensified follow-up schedule
  Interventions: Other: Intensified Follow-up Schedule
- B (Experimental): Adjuvant chemotherapy + intensified follow-up schedule
  Interventions: Drug: Capox (or FOLFOX) including flouropyrimidine and oxaliplatin combination chemotherapy

INTERVENTIONS:
Drug: Capox (or FOLFOX) including flouropyrimidine and oxaliplatin combination chemotherapy — Six months of adjuvant combination chemotherapy with Capox (or FOLFOX) Patients will receive adjuvant chemotherapy with eight cycles of CAPOX (oxaliplatin 130 mg/m2 day 1 and capecitabine 1000 mg/m2 b.i.d. days 1-14, repeated every 3 weeks.
  (Patients with an ileostomy are only eligible for FOLFOX and will be treated with 12 cycles of FOLFOX (oxaliplatin 85 mg/m2 day 1, leucovorin 400 mg/m2 day 1, 5FU 400 mg/m2 bolus day 1 and 5FU 2400 mg/ m2 over 46-48 hours day 1-3, repeated every second weeks)
  Arms: B
Other: Intensified Follow-up Schedule — Close monitoring with Imaging during follow-up Patients included in this trial will undergo intensified follow-up with CT-chest and abdomen every four months after surgery for the first 2 years, then every 6 months for 1 years and finally once yearly for the last 2 years up to 5 years follow-up is completed.
  Arms: A

SUMMARY:
A open label 1:1 randomized phase II exploratory study investigating adjuvant therapy in patients with molecular biologically detectable residual disease after primary resection for localized colorectal tumors.

DETAILED DESCRIPTION:
The main clinical hypothesis is that patients having undergone radical resection from CRC do not present with detectable tumor DNA in the plasma, whereas patients with detectable tumor DNA two weeks' post surgery have residual microscopic disease, and consequently a high risk of diseases recurrence which can be prevented with adjuvant chemotherapy.

The primary aim of the present study is to investigate - in a randomized trial - if use of standard adjuvant chemotherapy therapy improves the disease free survival in patients with molecular biological residual disease where adjuvant chemotherapy is not standard treatment .

Secondary aims include investigating molecular biological response to adjuvant chemotherapy in patients with post-operative ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Surgically removed Adenocarcinoma of the colon or rectum
* Pathologically stage I or II disease, and radical resection
* Detectable ctDNA in two weeks postoperative plasma sample
* No indication for adjuvant chemotherapy according to DCCG guidelines (website)
* Age at least 18 years
* ECOG performance status 0-2
* Clinically eligible for adjuvant chemotherapy at investigators decision.
* Adequate bone marrow, liver and renal function allowing systemic chemotherapy (Absolute neutrophil count ≥1.5x109/l and thrombocytes ≥ 100x109/l. Bilirubin ≤ 1.5 x upper normal value and alanine aminotransferase ≤ 3 x upper normal value, and Calculated or measured renal glomerular filtration rate at least 30 mL/min)
* Anticonception for fertile women and for male patients with a fertile partner. Intrauterine device, vasectomy of a female subject's male partner or hormonal contraceptive are acceptable •
* Written and verbally informed consent

Exclusion Criteria:

* Radiological evidence of distant metastasis, by CT- chest and abdomen
* Incapacity, frailty, disability and comorbidity to a degree that according to the investigator is not compatible with combination chemotherapy
* Previous treatment with 5FU or oxaliplatin
* Neuropathy NCI grade > 1
* Other malignant tumor within 5 years except non-melanoma skin cancer or carcinoma in situ cervicis uteri
* Pregnant (positive pregnancy test) or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
DFS | 3 years
  Disease free survival

SECONDARY OUTCOMES:
Molecular biological response | 6 months
  Molecular biological response at 6 months
MB-DFS | 1 year
  Molecular biological disease free survival at 1 year
TT-MBR | 3 years
  Time to molecular biological recurrence
TTR | 3 years
  Time to radiological recurrence
LRR | 3 years
  Local recurrence rate
DRR | 3 years
  Distant recurrence rate
OS | 5 years
  Overall survival
TR | 3 years
  Translational research exploratory

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No